CLINICAL TRIAL: NCT05449808
Title: Evaluation of the Appropriateness of Venous Thromboprophylaxis in Hospitalized Medical Patients Employing the Padua Prediction Score: an Observational Study
Brief Title: Evaluation of Thromboprophylaxis Appropriateness in Hospitalized Medical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al-Esraa University College (Other)
Responsible Party: Principal Investigator, Laith G. Shareef, Director, Al-Esraa University College
Other Study IDs: Venous thromboprophylaxis
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism; Venous Thromboses
Keywords: Padua prediction score; Pulmonary Embolism; Deep Vein Thrombosis; Venous Thromboses; Acute medical illness
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Considering observational studies that suggested a relationship between acutely ill medical patients and venous thromboembolism (VTE), interventional studies with anticoagulant medications indicated a marked decline in VTE during and after hospitalization. Despite the therapeutic value of lowering this result, there is a low inclination to utilize anticoagulants in patients hospitalized for acute medical diseases. This observational research aims to assess the appropriateness of venous thromboprophylaxis offered to patients admitted to internal medicine wards.

DETAILED DESCRIPTION:
Epidemiological studies have shown a significant prevalence of thromboembolism in patients admitted to medical wards.

Based on this, various clinical studies using anticoagulants such as unfractionated heparin (UFH), low-molecular-weight heparin (LMWH), and fondaparinux to prevent thromboembolism have been conducted in patients hospitalized for acute medical illness.

Interventional studies have repeatedly shown that anticoagulant prophylaxis lowers the incidence of deep venous thrombosis (DVT), pulmonary embolism (PE), and DVT-related mortality.

These findings led to recommendations to employ anticoagulant prophylaxis in patients hospitalized for acute medical disease; yet, anticoagulant prophylaxis is often underutilized in-hospital medical wards.

This study's primary objective is to assess the adequacy of venous thromboprophylaxis delivered to medical inpatients who need pharmacologic intervention in accordance with the American College of Chest Physicians (ACCP) guideline using the Padua prediction score.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Hospitalized for any cause in the internal medicine ward
* Ability to give informed consent, as informed by the physicians in charge of the patient

Exclusion Criteria:

* Expected hospital stay < 48 h
* Patients unable to give informed consent, as informed by the physicians in charge of the patient
* Patients with therapeutic anticoagulation at hospital admission
* Patients admitted for a disease requiring therapeutic anticoagulation
* Patients admitted to non-medical hospital wards

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Baghdad medical city; general internal medicine divisions patients'
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2022-11-13 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Appropriateness of venous thromboprophylaxis | August - December 2022
  The primary outcome of this study is to evaluate the appropriateness of venous thromboprophylaxis administered to medical inpatients who need pharmacologic interventions according to the American College of Chest Physicians (ACCP) 2012 guidelines and its second update in 2021.

SECONDARY OUTCOMES:
Reasons for insufficient venous thromboprophylaxis | August - December 2022
  The secondary purpose is to explore some significant reasons for insufficient venous thromboprophylaxis in various patients, such as prescription errors and administration mistakes.

CONTACTS AND LOCATIONS:
Overall Officials: Khulood M. Alsaraf, ASST PROF, Study Chair — Al-Esraa University College
Locations (1):
- EUC, Baghdad, Iraq

REFERENCES:
- [Background] Haas SK. Venous thromboembolic risk and its prevention in hospitalized medical patients. Semin Thromb Hemost. 2002 Dec;28(6):577-84. doi: 10.1055/s-2002-36702. PMID 12536351
- [Background] Barbar S, Noventa F, Rossetto V, Ferrari A, Brandolin B, Perlati M, De Bon E, Tormene D, Pagnan A, Prandoni P. A risk assessment model for the identification of hospitalized medical patients at risk for venous thromboembolism: the Padua Prediction Score. J Thromb Haemost. 2010 Nov;8(11):2450-7. doi: 10.1111/j.1538-7836.2010.04044.x. PMID 20738765